CLINICAL TRIAL: NCT01105013
Title: Study Clinical, Multicenter, Phase III, to Evaluate the Efficacy and Safety of Tolnaftate Cream in the Treatment of Patients With Fungal Infections Like Tinea Foot, Tinea and Tinea Crural Body"
Brief Title: Evaluate the Efficacy and Safety of Tolnaftate Cream in the Treatment of Patients With Fungal Infections
Acronym: Tonaftato
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratório Teuto Brasileiro S/A (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEU-TOL-03/09
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Fungal Infections; Tinea Pedis; Tinea Cruris; Tinea Corporis
Keywords: fungal infections; tinea; tonaftato
MeSH Terms: conditions — Mycoses; Tinea Pedis; Tinea Cruris; Tinea | interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tonaftato (Experimental): Apply the product in sufficient quantity to cover the affected area 2 times daily (every 12 hours) for 60 days.
  Interventions: Drug: Clotrimazole

INTERVENTIONS:
Drug: Clotrimazole — Apply the product in sufficient quantity to cover the affected area 2 times daily (every 12 hours) for 60 days.

SUMMARY:
This is a study clinical, multicenter, Phase III trial, to evaluate the efficacy and safety of tolnaftate cream in the treatment of patients with fungal infections such as Tinea foot, Tinea and Tinea crural body.

DETAILED DESCRIPTION:
Study Clinical, multicenter, Phase III, to evaluate the efficacy and safety of 10mg/g tolnaftate cream in the treatment of patients with fungal infections such as Tinea foot, Tinea and Tinea crural body.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, of any race, aged 12 years;
* Ability to understand and sign the IC (for patients older than age) in the case of minors monitoring and consent of a guardian;
* Clinical diagnosis of fungal infections for tinea pedis (ringworm of the feet) or tinea cruris (ringworm of the groin region), or tinea corporis (ringworm in other body areas);
* Direct mycological exam positive for fungi;

Exclusion Criteria:

* Pregnant women or nursing mothers;
* Use of topical or oral antifungal;
* Use of steroids;
* Allergy or hypersensitivity to any component of product;
* Clinical cases of tinea infection by bacteria and / or eczema, tinea extensive and onychomycosis.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy and safety of the tolnaftate cream 10 mg / g. | 97 days
  Apply the product in sufficient quantity to cover the affected area 2 times daily (every 12 hours) for 60 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dagoberto Brandão, Study Director — PHC - Pharma Consulting
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil